CLINICAL TRIAL: NCT01270828
Title: A Phase 3 Double-blind, Randomized, Placebo-controlled, Safety And Efficacy Study Of Once Daily Controlled Release Pregabalin In The Treatment Of Patients With Postherpetic Neuralgia (Protocol A0081224)
Brief Title: Safety And Efficacy Study Of Once Daily Controlled Release Pregabalin In The Treatment Of Patients With Postherpetic Neuralgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081224; 2009-016766-86 (EudraCT Number)
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Results first posted 2016-01-13 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2015-12

CONDITIONS: Post Herpetic Neuralgia
Keywords: Control Release Pregabalin in Post Herpetic Neuralgia
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pregablain CR tablet 82.5 to 660mg (Experimental)
  Interventions: Drug: Pregabalin
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Pregabalin — Tablets, 82.5 to 660mg, once per day. Duration: 19 weeks
  Arms: Pregablain CR tablet 82.5 to 660mg
Drug: placebo — Placebo, 82.5 to 660mg, once per day. Duration: 13 weeks
  Arms: Placebo

SUMMARY:
The purpose of the study is to explore the safety and efficacy of a new once a day pregabalin formulation versus placebo for patients with post herpetic neuralgia (Shingles)

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pain present for more than 3 months after the healing of the herpes zoster skin rash.
* At screening (V1) and enrollment (V2), patients must have a score of greater than or equal to 4 on the Pain Numeric Rating Scale (1 week recall period).
* At enrollment (V2), at least 4 pain diaries must be completed satisfactorily within the last 7 days and the average pain score must be greater than or equal to 4.
* Male or female of any race, at least 18 years of age, and using appropriate methods of contraception

Exclusion Criteria:

* Creatinine clearance <30 mL/min (estimated from serum creatinine).
* Skin conditions in the affected dermatome that could alter sensation
* Pregabalin use in the last 30 days. Subjects taking pregabalin in the last 30 days should be washed out of pregabalin for at least 30 days prior to screening visit. Patients who had not responded to pregabalin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 806 (Actual)
Dates: Start 2011-03; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (144):
- United States (81):
  - Fundamental Research, Gulf Shores, Alabama
  - Radiant Research, Inc., Chandler, Arizona
  - Elite Clinical Studies, LLC, Phoenix, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - The Pain Center of Arizona, Phoenix, Arizona
  - Genova Clinical Research, Tucson, Arizona
  - Larry Watkins, M.D. (Private Practice), Little Rock, Arkansas
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Hearne Family Practice Clinic, Little Rock, Arkansas
  - Center for Clinical Research, Inc, Carmichael, California
  - Community Medical Providers, Clovis, California
  - Sierra Medical Research, Clovis, California
  - Inland Pain Medicine, Colton, California
  - The Helm Center, Laguna Hills, California
  - University of Southern California, Los Angeles, California
  - USC IDS Pharmacy, Los Angeles, California
  - Translational Research Group, Inc, North Hollywood, California
  - George J. Rederich, M.D., Incorporated, Redondo Beach, California
  - Integrated Research Group, Inc., Riverside, California
  - Drug Shipmnent Only Aristotelis T. Laliotis, M.D. Integrated Research Center, Inc., San Diego, California
  - Integrated Research Center, Inc., San Diego, California
  - Center For Clinical Research, Inc., San Francisco, California
  - Neurological Research Institute, Santa Monica, California
  - Foothills Pain Management Clinic, PS, West Covina, California
  - JEM Research Institute, Atlantis, Florida
  - Orthopedic Research Institute, Boynton Beach, Florida
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Clinical Physiology Associates, Fort Myers, Florida
  - Health Care Family Rehab & Research Center, Hialeah, Florida
  - Laszlo Jozsef Mate, MD, North Palm Beach, Florida
  - Family Care Specialists, Ocala, Florida
  - Renstar Medical Research, Ocala, Florida
  - Compass Research, LLC, Orlando, Florida
  - Comprehensive Pain care of South Florida, Royal Palm Beach, Florida
  - Comprehensive Clinical Development Inc., St. Petersburg, Florida
  - Neurology Clinical Research, Inc., Sunrise, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Meridien Research, Tampa, Florida
  - Injury Care Medical Center, Boise, Idaho
  - Millennium Pain Center, LLC, Bloomington, Illinois
  - (IP Shipping Address) Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Chicago Anesthesia Pain Specialists, Chicago, Illinois
  - Advanced Pain Care Clinic, Evansville, Indiana
  - Clinical Research Advantage, Evansville, Indiana
  - Global Scientific Innovations, Evansville, Indiana
  - Clinical Trials of America, Inc., Monroe, Louisiana
  - Boston Clinical Trials, Boston, Massachusetts
  - Beacon Clinical Research, Brockton, Massachusetts
  - Infinity Medical Research, Inc., North Dartmouth, Massachusetts
  - Michigan Head Pain & Neurological Institute, Ann Arbor, Michigan
  - QUEST Research Institute, Bingham Farms, Michigan
  - The Center for Pharmaceutical Research, PC, Kansas City, Missouri
  - Clinvest, A Division of Banyan Group, Inc, Springfield, Missouri
  - Medex Healthcare Research, Inc., St Louis, Missouri
  - Montana Medical Research Inc, Missoula, Montana
  - Lincoln Internal Medicine Associates, Lincoln, Nebraska
  - Drug Shipment Only: Heartland Clinical Research, Inc., Omaha, Nebraska
  - Heartland Clinical Research, Inc., Omaha, Nebraska
  - The Office of Dr. Stephen H. Miller, MD, Las Vegas, Nevada
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Dent Neurological Institute, Amherst, New York
  - SPRI Clinical Trials LLC, Brooklyn, New York
  - Medex Healthcare Research, Inc - Saint Louis, New York, New York
  - North American Partners In Pain Management, New York, New York
  - Asheville Neurology Specialists, PA, Asheville, North Carolina
  - Raleigh Neurology Associates, P.A., Raleigh, North Carolina
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Radiant Research, Akron, Ohio
  - Providence Health Partners-Center for Clinical Research, Dayton, Ohio
  - Wells Institute for Health Awareness, Kettering, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Mark A Fisher, Oklahoma City, Oklahoma
  - Pharmacorp Clinical Trials, Inc., Charleston, South Carolina
  - Arlington Research Center, Inc., Arlington, Texas
  - Lovelace Scientific Resources, Inc., Austin, Texas
  - Radiant Research, Dallas, Texas
  - ClinRx Research, LLC, Richardson, Texas
  - Hillcrest Family Health Centers, Division of Clinical Research, Waco, Texas
  - Clinical Research Associates of Tidewater, Norfolk, Virginia
  - Clinical Investigation Specialists, Inc., Kenosha, Wisconsin
- Bulgaria (6):
  - DCC "St. Pantaleimon" OOD, Pleven
  - MHAT-Pleven, Pleven
  - MBALNP "Sveti Naum" EAD, Klinika po nervni bolesti za dvigatelni narushenia, Sofia
  - Vtora Mnogoprofilna Bolnitsa za Aktivno Lechenie ¿ Sofia, AD, Sofia, Nevrologichno otdelenie, Sofia
  - MBAL "Tokuda Bolnitsa", Otdelenie po nevrologiya, Sofia
  - Universitetska mnogoprofilna bolnitsa za aktivno lechenie Aleksandrovska, Klinika po Nevrologia, Sofia
- Colombia (3):
  - Reumalab S.A.S, Medellín, Antioquia
  - Centro de Investigacion y Atencion Para la Salud Mental S.A. - CESAME, Bogota, Cundinamarca
  - Fundacion Cardiovascular de Colombia, Floridablanca, Santander Department
- Croatia (3):
  - Opca bolnica Karlovac, Karlovac, Karlovacka Županija
  - Klinicki Bolnicki Centar Osijek, Osijek, Osjecko-baranjska Županija
  - Opca bolnica "Dr. Ivo Pedisic", Sisak, Sisacko-moslavacka Županija
- Neurologicka ambulance, Prerov I, Czechia
- Denmark (2):
  - Aalborg Sygehus Nord, Aalborg, North Denmark
  - Glostrup Hospital, Glostrup Municipality
- Germany (3):
  - Schmerzzentrum Frankfurt, Frankfurt am Main, Hesse
  - pro scientia med im MARE Klinikum, Kiel-Kronshagen, Schleswig-Holstein
  - DGS-Schmerzzentrum Eichstätt, Eichstätt
- Hong Kong (2):
  - Family Medicine, Hong Kong
  - Queen Elizabeth Hospital, Kowloon
- India (5):
  - Medanta Institute of Neurosciences, Gurgaon, Haryana
  - Manipal Hospital, Bangalore, Karnataka
  - M. S. Ramaiah Medical College and Hospitals, Bangalore, Karnataka
  - Mallikatta Neuro Centre, Mangalore, Karnataka
  - Indraprastha Apollo Hospitals, New Delhi
- Poland (6):
  - "SYNEXUS POLSKA" Sp. z o.o., Wroclaw, Lower Silesian Voivodeship
  - Prof. dr hab. med. Leszek Szepanski Prywatna Praktyka Lekarska Gabinet Reumatologiczny, Lublin, Lublin Voivodeship
  - "SYNEXUS POLSKA" Sp. z o.o. Oddzial w Warszawie, Warsaw, Masovian Voivodeship
  - Niepubliczny Zaklad Opieki Zdrowotnej "Przychodnia Morena" Sp. z o.o., Gdansk, Pomeranian Voivodeship
  - "SYNEXUS POLSKA" Sp. z o.o. Oddzial w Gdyni, Gdynia, Pomeranian Voivodeship
  - "SYNEXUS POLSKA" Sp. z o.o. Oddzial w Katowicach, Katowice, Silesian Voivodeship
- Russia (7):
  - State Budgetary Health Institution of Yaroslavl region "Clinical hospital #10", Yaroslavl, Russian Federation
  - State Budgetary Educational Institution for higher Professional Training "Kazan State Medical Univer, Kazan', Tatarstan, Respublika
  - Kazan State Medical University, Kazan', Tatarstan, Respublika
  - GBUZ Nizhny Novgorod Regional Clinical Hospital N.A. Semashko, Nizhny Novgorod
  - Clinic of Nervous Diseases M.I. Astvatsaturov, Saint Petersburg
  - St. Petersburg State Healthcare Institution City Hospital # 40 Kurortnogo Administrativnogo Rajona, Saint Petersburg
  - State Budgetary Educational Institution for Higher Professional Education, Smolensk
- Serbia (2):
  - Clinic for Neurology, Belgrade
  - Clinic for Neurology, Niš
- Slovakia (4):
  - Euro-Neuro s.r.o., Neurologicka ambulancia, Bratislava
  - Univerzitna nemocnica Bratislava, Nemocnica sv. Cyrila a Metoda, Neurologicke oddelenie, Bratislava
  - MUDr. Eva Gasparova - neurologicka ambulancia, Hlohovec
  - Neurologicka ambulancia, Neuron-DT,s.r.o., Žilina
- South Africa (5):
  - Nelson Mandela Academic Hospital Research Unit, Mthatha, Eastern Cape
  - Iatros International, Bloemfontein
  - Synapta Clinical Research Centre, Durban
  - Mzansi Ethical Research Centre, Middelburg
  - Jakaranda Pain Clinic, Pretoria
- Sweden (5):
  - Probare, Lund, Skåne County
  - Me3plus Clinical Trials, Gothenburg
  - CTC, Sahlgrenska sjukhuset/SU, Gothenburg
  - Center for Lakemedelsstudier, Malmo
  - Bragee Medect AB, Stockholm
- Taiwan (2):
  - Chang Gung Medical Foundation-Linkou Branch, Kwei Shan Town, Taoyuan County
  - National Taiwan University Hospital (Neurology), Taipei
- Ukraine (7):
  - Public Institution "Institute of Neurology, Psychiatry and Narcology of AMS of Ukraine", Kharkiv
  - Kyiv City Clinical Hospital #4, Kyiv
  - Lviv NMU n.a. Danylo Galytskyy, Lviv
  - Regional Municipal Dermatovenerologic Dispensary, Lviv
  - Crimean Republican Institution "Clinical Dermatovenerologic Dispensary", Simferopol
  - Municipal Establishment "Vinnitsa Regional Psychoneurological Hospital n.a. O.I. Yushchenko", Vinnitsa
  - Municipal Establishment "City Clinical Hospital #2", Neurology Department, Zaporizhzhya

REFERENCES:
- [Derived] Huffman CL, Goldenberg JN, Weintraub J, Sanin L, Driscoll J, Yang R, Chew ML, Scavone JM. Efficacy and Safety of Once-Daily Controlled-Release Pregabalin for the Treatment of Patients With Postherpetic Neuralgia: A Double-Blind, Enriched Enrollment Randomized Withdrawal, Placebo-Controlled Trial. Clin J Pain. 2017 Jul;33(7):569-578. doi: 10.1097/AJP.0000000000000445. PMID 27753650
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081224&StudyName=Safety%20And%20Efficacy%20Study%20Of%20Once%20Daily%20Controlled%20Release%20Pregabalin%20In%20The%20Treatment%20Of%20Patients%20With%20Postherpetic%20Neuralgia%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 129 centers in 17 countries screened subjects for the study, including 68 in the US, 6 in Bulgaria, 6 in Poland, 6 in Russia, 6 in the Ukraine, 5 in India, 5 in South Africa, 5 in Sweden, 4 in Slovakia, 3 in Colombia, 3 in Croatia, 3 in Germany, 2 in Denmark, 2 in Hong Kong, 2 in Serbia, 2 in Taiwan, and 1 in the Czech Republic.
Pre-assignment Details: The study consisted of 4 phases: Baseline (1 week [wk]): to determine study entry criteria; Single Blind (SB) (6 wks): to determine optimized dose; Double Blind (DB) (13 wks): responders with at least 50% improvement in pain at SB were considered and randomized to pregabalin or matching placebo; and DB taper phase (1 wk).
Groups:
- Pregabalin Controlled Release (CR) DB: Possible doses for participants with normal creatinine clearance (CLcr) (≥60 mL/min) during the DB fixed dose phase were pregabalin CR 165 mg/day, 330 mg/day, 495 mg/day CR or 660 mg/day CR. Doses for participants with low CLcr (>30 - <60 mL/min) were pregabalin 82.5 mg/day, 165 mg/day, 247.5 mg/day, or 330 mg/day CR.
- Placebo DB: Participants received matching placebo
- Pregabalin CR SB: The participants with normal CLcr (≥60 mL/min) were treated with pregabalin 165 mg/day CR; those with low CLcr (>30 - <60 mL/min) received 82.5 mg/day pregabalin CR. Subsequently, the pregabalin doses were increased based on efficacy and tolerability at each weekly visit.
Period: Pregabalin CR SB
Arm/Group | Pregabalin Controlled Release (CR) DB | Placebo DB | Pregabalin CR SB
Started | 0 | 0 | 806
Completed | 0 | 0 | 660
Not Completed | 0 | 0 | 146
Not completed — Reason Unspecified | 0 | 0 | 8
Not completed — Enrolled but not treated | 0 | 0 | 5
Not completed — Related adverse event | 0 | 0 | 46
Not completed — Lack of Efficacy | 0 | 0 | 32
Not completed — Withdrawal by Subject | 0 | 0 | 29
Not completed — Lost to Follow-up | 0 | 0 | 10
Not completed — Unrelated AE | 0 | 0 | 8
Not completed — Protocol Violation | 0 | 0 | 8
Period: Double Blind Phase
Arm/Group | Pregabalin Controlled Release (CR) DB | Placebo DB | Pregabalin CR SB
Started | 208 | 205 | 0
Completed | 182 | 160 | 0
Not Completed | 26 | 45 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Protocol and GCP non-compliance | 4 | 3 | 0
Not completed — Reason Unspecified | 7 | 4 | 0
Not completed — Withdrawal by Subject | 6 | 15 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0
Not completed — Lack of Efficacy | 2 | 11 | 0
Not completed — Adverse event not related to study drug | 1 | 1 | 0
Not completed — Adverse event related to study drug | 5 | 7 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population description consisted of all participants randomized to the DB phase who received at least 1 dose of study medication in the DB phase (full analysis set).
Groups:
- Pregabalin CR DB: Possible doses for participants with normal creatinine clearance (CLcr) (≥60 mL/min) during the DB fixed dose phase were pregabalin CR 165 mg/day, 330 mg/day, 495 mg/day CR or 660 mg/day CR. Doses for participants with low CLcr (>30 - <60 mL/min) were pregabalin 82.5 mg/day, 165 mg/day, 247.5 mg/day, or 330 mg/day CR.
- Total: Total of all reporting groups
Arm/Group | Pregabalin CR DB | Placebo DB | Total
Number analyzed (Participants) | 208 | 205 | 413
Age, Customized [Number; unit: Participants]
  <18 years | 0 | 0 | 0
  18-44 years | 26 | 24 | 50
  45-64 years | 86 | 78 | 164
  ≥65 years | 96 | 103 | 199
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 122 | 256
  Male | 74 | 83 | 157

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Loss of Therapeutic Response.
Description: Loss of Therapeutic Response (LTR) is defined as <30% pain response relative to the single blind phase baseline or patient discontinuation due to lack of efficacy or adverse events in the double blind phase of the study. For the calculation of <30% pain response relative to baseline, baseline will be defined as the mean of the last 7 observations prior to the start of SB treatment, which will be compared with the 7 days rolling average of pain response in DB phase. Participants may be discontinued due to lack of efficacy in this study at the discretion of the study physician.
Time Frame: 13 Weeks
Population: The full analysis set (FAS) was the primary efficacy analysis set and consisted of all participants randomized to the DB phase who received at least 1 dose of study drug in the DB phase.
Measure: Number; unit: Participants
Arm/Group | Pregabalin CR DB | Placebo DB
Number analyzed (Participants) | 208 | 205
Participants | 29 | 63
Statistical Analysis 1: Comparison: Pregabalin CR DB vs Placebo DB; Kaplan-Meier method was used for the analysis; Test type: Superiority or Other; p < 0.0001, Log Rank

2. Secondary Outcome: Participants With Secondary LTR Based on 5 Day Rolling Average Diary Results
Description: A secondary LTR endpoint (S-LTR) was defined as the 5 day rolling average pain score during DB, compared to the 5 day randomization baseline pain score. As a secondary endpoint, S-LTR was defined as:
  1. At least a 30% increase in the 5 days rolling average pain score during DB relative to the 5 Day randomization baseline pain score
  2. A 5 days rolling average pain score ≥4. Participants who discontinue due to lack of efficacy or adverse events in the DB phase of the study will also be counted as an LTR.
Time Frame: 13 Weeks
Population: The FAS consisted of all participants randomized to the DB phase who received at least 1 dose of study drug in the DB phase
Measure: Number; unit: Participants
Arm/Group | Pregabalin CR DB | Placebo DB
Number analyzed (Participants) | 208 | 205
Participants | 49 | 87
Statistical Analysis 1: Comparison: Pregabalin CR DB vs Placebo DB; Kaplan-Meier method was used for the analysis; Test type: Superiority or Other; p < 0.0001, Log Rank

3. Secondary Outcome: Percentage of Participants With 30% Reduction in the Mean Pain Score.
Description: The 30% pain responders were defined as participants with at least a 30% reduction in the mean pain score from SB baseline to DB endpoint.
Time Frame: 13 Weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin CR DB | Placebo DB
Number analyzed (Participants) | 206 | 204
Percentage of participants | 95.6 | 83.8
Statistical Analysis 1: Comparison: Pregabalin CR DB vs Placebo DB; Chi-square test was used for analysis; Test type: Superiority or Other; p < 0.0001, Chi-squared

4. Secondary Outcome: Percentage of Participants With 50% Reduction in the Mean Pain Score.
Description: The 50% pain responders were defined as participants with at least a 50% reduction in the mean pain score from SB baseline to DB endpoint.
Time Frame: 13 Weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin CR DB | Placebo DB
Number analyzed (Participants) | 206 | 204
Percentage of participants | 88.3 | 68.6
Statistical Analysis 1: Comparison: Pregabalin CR DB vs Placebo DB; Chi-square test was used for analysis; Test type: Superiority or Other; p < 0.0001, Chi-squared

5. Secondary Outcome: Change From Baseline to Endpoint in Weekly Mean Pain Score.
Description: The pain numeric rating scale (NRS Pain) consists of an 11 point NRS ranging from 0 (no pain) to 10 (worst possible pain). A rating of 1-3 is considered mild pain; 4-6, moderate pain; and 7-10, severe pain
Time Frame: SB Baseline (Enrollment) to Week 19 and DB Baseline (Week 6) to Week 19
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin CR DB | Placebo DB
Number analyzed (Participants) | 206 | 205
Units on a scale
  SB Baseline to Week 19 | -4.89 (0.12) | -3.95 (0.12)
  DB Baseline to Week 19 | -0.04 (0.11) | 0.87 (0.11)
Statistical Analysis 1: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for SB Baseline to Week 19. Estimates and p-values are from an ANCOVA main effects model with baseline value, pooled center decided before unblinding, and treatment in the model; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.94, 95% CI 2-sided [-1.26 to -0.62], Standard Error of Mean 0.16
Statistical Analysis 2: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for DB Baseline to Week 19. Estimates and p-values are from an ANCOVA main effects model with baseline value, pooled center decided before unblinding, and treatment in the model; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.91, 95% CI 2-sided [-1.21 to -0.61], Standard Error of Mean 0.15

6. Secondary Outcome: Change in the Weekly NRS-Pain (1-Week Recall).
Description: The pain numeric rating scale (NRS Pain) consists of an 11 point NRS ranging from 0 (no pain) to 10 (worst possible pain). A rating of 1-3 is considered mild pain; 4-6, moderate pain; and 7-10, severe pain. Participants were asked to rate their pain over the past week.
Time Frame: SB Baseline (Enrollment) to Week 19 and DB Baseline (Week 6) to Week 19
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin CR DB | Placebo DB
Number analyzed (Participants) | 203 | 195
Units on a scale
  SB Baseline to Week 19 | -5.0 (0.13) | -3.9 (0.14)
  DB Baseline to Week 19 | -0.1 (0.13) | 0.9 (0.13)
Statistical Analysis 1: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for SB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-1.47 to -0.75]
Statistical Analysis 2: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for DB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-1.34 to -0.65]

7. Secondary Outcome: Change in the Medical Outcomes Study-Sleep Scale (MOS-SS).
Description: The MOS-SS is a validated self administered questionnaire consisting of 12 items that assess key constructs of sleep. The scale has been found reliable and valid with good overall measurement properties. Instrument scoring yields 7 subscales (sleep disturbance, snoring, awaken short of breath or with a headache, quantity of sleep, optimal sleep, sleep adequacy, and somnolence) as well as a 9 item overall sleep problems index assessing sleep over the past week. Scores are transformed (actual raw score minus lowest possible score divided by possible raw score range multiplied by 100); total score range = 0 to 100; higher score indicates greater intensity of attribute.
Time Frame: SB Baseline (BL) (Enrollment) to Week 19 and DB Baseline (Week 6) to Week 19
Population: The FAS consisted of all participants randomized to the DB phase who received at least 1 dose of study drug in the DB phase. N in the below table refers to number of participants analyzed: 203 in Pregabalin DB CR group and 195 in Placebo DB group, unless otherwise specified.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin CR DB | Placebo DB
Number analyzed (Participants) | 203 | 195
Units on a scale
  Sleep Problems Index I-SB BL to wk 19(N=202,195) | -19.9 (1.09) | -16.7 (1.13)
  Sleep Problems Index I-DB BL to wk 19(N=202,195) | 1.2 (1.05) | 4.4 (1.09)
  SleepProblems Index II-SB BL to wk 19(N=202,195) | -21.2 (1.07) | -17.4 (1.11)
  SleepProblems Index II-DB BL to wk 19(N=202,194) | 0.2 (1.01) | 4.3 (1.05)
  Sleep Disturbance-SB BL to wk 19 | -28.3 (1.42) | -21.1 (1.48)
  Sleep Disturbance-DB BL to wk 19 | -1.1 (1.31) | 7.6 (1.36)
  Snoring-SB BL to wk 19(N=202,194) | -3.3 (1.57) | -4.7 (1.64)
  Snoring-DB BL to wk 19(N=201,194) | -0.6 (1.41) | 0.8 (1.46)
  Awaken short of breath/headache-SB BL to wk 19 | -11.9 (1.21) | -10.4 (1.26)
  Awaken short of breath/headache-DB BL to wk 19 | -1.2 (1.23) | -0.2 (1.27)
  Sleep adequacy-SB BL to wk 19 | 19.9 (1.83) | 17.5 (1.90)
  Sleep adequacy-DB BL to wk 19(N=202,195) | -3.3 (1.82) | -6.0 (1.89)
  Somnolence-SB BL to wk 19(N=202,195) | -12.0 (1.19) | -12.0 (1.23)
  Somnolence-DB BL to wk 19(N=203,194) | -0.7 (1.15) | -0.9 (1.19)
Statistical Analysis 1: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Sleep Problem Index I-SB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.0324, ANCOVA; Mean Difference (Final Values) = -3.2, 95% CI 2-sided [-6.1 to -0.3]
Statistical Analysis 2: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Sleep Problem Index I-DB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.0223, ANCOVA; Mean Difference (Final Values) = -3.3, 95% CI 2-sided [-6.1 to -0.5]
Statistical Analysis 3: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Sleep Problem Index II-SB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.0098, ANCOVA; Mean Difference (Final Values) = -3.8, 95% CI 2-sided [-6.6 to -0.9]
Statistical Analysis 4: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Sleep Problem Index II-DB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.0033, ANCOVA; Mean Difference (Final Values) = -4.0, 95% CI 2-sided [-6.7 to -1.4]
Statistical Analysis 5: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Sleep Disturbance-SB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.0002, ANCOVA; Mean Difference (Final Values) = -7.3, 95% CI 2-sided [-11.1 to -3.5]
Statistical Analysis 6: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Sleep Disturbance-DB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -8.7, 95% CI 2-sided [-12.2 to -5.2]
Statistical Analysis 7: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Snoring-SB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.5264, ANCOVA; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [-2.8 to 5.6]
Statistical Analysis 8: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Snoring-DB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.4520, ANCOVA; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-5.2 to 2.3]
Statistical Analysis 9: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Awaken Short of Breath or with a Headache-SB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.3714, ANCOVA; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-4.7 to 1.8]
Statistical Analysis 10: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Awaken Short of Breath or with a Headache-DB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.5639, ANCOVA; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-4.2 to 2.3]
Statistical Analysis 11: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Sleep adequacy-SB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.3223, ANCOVA; Mean Difference (Final Values) = 2.5, 95% CI 2-sided [-2.4 to 7.3]
Statistical Analysis 12: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Sleep adequacy-DB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.2742, ANCOVA; Mean Difference (Final Values) = 2.7, 95% CI 2-sided [-2.2 to 7.6]
Statistical Analysis 13: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Somnolence-SB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.9816, ANCOVA; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-3.2 to 3.1]
Statistical Analysis 14: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Somnolence-DB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.9282, ANCOVA; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-2.9 to 3.2]

8. Secondary Outcome: Change in the MOS-SS-Quantity of Sleep.
Description: The MOS-SS is a validated self administered questionnaire consisting of 12 items that assess key constructs of sleep. The scale has been found reliable and valid with good overall measurement properties. Instrument scoring yields 7 subscales (sleep disturbance, snoring, awaken short of breath or with a headache, quantity of sleep, optimal sleep, sleep adequacy, and somnolence) as well as a 9 item overall sleep problems index assessing sleep over the past week.
  The item "Quantity of sleep" of MOS-SS is presented here.
Time Frame: SB Baseline (BL) (Enrollment) to Week 19 and DB Baseline (Week 6) to Week 19
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | Pregabalin CR DB | Placebo DB
Number analyzed (Participants) | 203 | 192
Hours
  Quantity of sleep-SB BL to wk 19(N=203,192) | 0.9 (0.09) | 0.7 (0.10)
  Quantity of sleep-DB BL to wk 19(N=202,192) | -0.1 (0.08) | -0.4 (0.09)
Statistical Analysis 1: Comparison: Pregabalin CR DB vs Placebo DB; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.1635, ANCOVA; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.1 to 0.4]
Statistical Analysis 2: Comparison: Pregabalin CR DB vs Placebo DB; [analysis description as in outcome 6, analysis 2]; Test type: Superiority or Other; p = 0.0363, ANCOVA; Mean Difference (Final Values) = 0.2, 95% CI [0.0 to 0.5]

9. Secondary Outcome: The MOS-SS-Optimal Sleep.
Description: The MOS-SS is a validated self administered questionnaire consisting of 12 items that assess key constructs of sleep. The scale has been found reliable and valid with good overall measurement properties. Instrument scoring yields 7 subscales (sleep disturbance, snoring, awaken short of breath or with a headache, quantity of sleep, optimal sleep, sleep adequacy, and somnolence) as well as a 9 item overall sleep problems index assessing sleep over the past week.
  The optimal sleep score is a dichotomous 'Yes' or 'No' rating, where 'Yes' indicates optimal sleep (average 7-8 hours per night) and 'No' indicates not optimal sleep. The "percentage of participants with optimal sleep" is presented here.
Time Frame: Week 6 and Week 19
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin CR DB | Placebo DB
Number analyzed (Participants) | 208 | 205
Percentage of participants
  Week 6 (N=208,205) | 58.7 (0.09) | 62.4 (0.10)
  Week 19 (N=204,197) | 54.9 (0.08) | 54.8 (0.09)
Statistical Analysis 1: Comparison: Pregabalin CR DB vs Placebo DB; This analysis is for Week 6; Test type: Superiority or Other; p = 0.432, Chi-squared
Statistical Analysis 2: Comparison: Pregabalin CR DB vs Placebo DB; This analysis is for Week 19; Test type: Superiority or Other; p = 0.987, Chi-squared

10. Secondary Outcome: Percentage of Participants With Change in the Patient Global Impression of Change (PGIC) Score
Description: The PGIC is a participant-rated instrument that has been used in chronic pain and fibromyalgia studies to rate change in a patient's overall status. This single item instrument uses a 7 point Likert scale, anchored by (1) very much improved, to (7) very much worse.
Time Frame: Week 19
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin CR DB | Placebo DB
Number analyzed (Participants) | 203 | 195
Percentage of participants
  Very much improved | 31.5 | 23.1
  Much improved | 36.9 | 30.3
  Minimally improved | 16.7 | 19.0
  No change | 10.3 | 12.8
  Minimally worse | 2.5 | 7.2
  Much worse | 1.5 | 7.2
  Very much worse | 0.5 | 0.5
Statistical Analysis 1: Comparison: Pregabalin CR DB vs Placebo DB; This analysis is for the original score. Proportional odds Logistic regression with a term for treatment in the model; Test type: Superiority or Other; p = 0.0007, Regression, Logistic; Odds Ratio (OR) = 1.85, 95% CI 2-sided [1.30 to 2.65] — Odds ratio is the probability of the event occurring in Pregabalin DB relative to the event occurring in Placebo DB. Odds ratio > 1 is in favor of Pregabalin DB
Statistical Analysis 2: Comparison: Pregabalin CR DB vs Placebo DB; This analysis is for the categorized score. Proportional odds Logistic regression with a term for treatment in the model; Test type: Superiority or Other; p = 0.0009, Regression, Logistic; Odds Ratio (OR) = 2.32, 95% CI 2-sided [1.41 to 3.81] — [estimate comment as in outcome 10, analysis 1]

11. Secondary Outcome: Change in the Short Form 36 Health Survey (SF-36)
Description: The SF 36 is a self administered, validated questionnaire that measures each of the following 8 health aspects: Physical functioning, role limitations due to physical problems, social functioning, bodily pain, mental health, role limitations due to emotional problems, vitality, and general health perception over the past week. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning) where, higher scores indicate a better health related quality of life.
Time Frame: Week 19
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin CR DB | Placebo DB
Number analyzed (Participants) | 203 | 195
Units on a scale
  Physical Component-SB BL to wk 19(N=202,195) | 7.5 (0.54) | 5.6 (0.56)
  Physical Component-DB BL to wk 19(N=202,195) | 0.1 (0.51) | -2.3 (0.53)
  Mental Component-SB BL to wk 19(N=202,195) | 6.4 (0.62) | 5.5 (0.64)
  Mental Component-DB BL to wk 19(N=202,195) | -1.1 (0.62) | -2.2 (0.64)
  Physical functioning-SB BL to wk 19 | 11.7 (1.44) | 8.9 (1.49)
  Physical functioning-DB BL to wk 19 | -1.4 (1.25) | -4.9 (1.29)
  Role-Physical-SB BL to wk 19 | 18.9 (1.62) | 13.9 (1.67)
  Role-Physical-DB BL to wk 19 | -2.4 (1.54) | -7.7 (1.60)
  Bodily pain-SB BL to wk 19 | 31.0 (1.51) | 23.6 (1.56)
  Bodily pain-DB BL to wk 19 | 1.4 (1.38) | -6.2 (1.43)
  General Health Perception-SB BL to wk19(N=202,195) | 11.3 (1.05) | 8.2 (1.08)
  General Health Perception-DB BL to wk19(N=202,195) | 1.4 (0.96) | -4.0 (1.00)
  Vitality-SB BL to wk 19(N=202,195) | 13.7 (1.25) | 10.7 (1.30)
  Vitality-DB BL to wk 19(N=202,195) | -3.5 (1.21) | -6.5 (1.25)
  Social Functioning-SB BL to wk 19 | 18.5 (1.35) | 15.7 (1.39)
  Social Functioning-DB BL to wk 19 | -2.1 (1.28) | -4.3 (1.32)
  Role-Emotional-SB BL to wk 19 | 15.0 (1.43) | 11.6 (1.47)
  Role-Emotional-DB BL to wk 19 | -1.4 (1.42) | -5.4 (1.47)
  Mental Health-SB BL to wk 19(N=202,195) | 11.1 (1.05) | 9.5 (1.08)
  Mental Health-DB BL to wk 19(N=202,195) | -1.3 (1.04) | -3.7 (1.08)
Statistical Analysis 1: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Bodily pain-SB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.0003, ANCOVA; Mean Difference (Final Values) = 7.4, 95% CI 2-sided [3.4 to 11.5]
Statistical Analysis 2: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Bodily pain-DB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 7.7, 95% CI 2-sided [4.0 to 11.3]
Statistical Analysis 3: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for General Health Perceptions-SB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.0275, ANCOVA; Mean Difference (Final Values) = 3.2, 95% CI 2-sided [0.4 to 6.0]
Statistical Analysis 4: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for General Health Perceptions-DB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 5.4, 95% CI 2-sided [2.8 to 8.0]
Statistical Analysis 5: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Vitality-SB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.0735, ANCOVA; Mean Difference (Final Values) = 3.0, 95% CI 2-sided [-0.3 to 6.4]
Statistical Analysis 6: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Vitality-DB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.0684, ANCOVA; Mean Difference (Final Values) = 3.0, 95% CI 2-sided [-0.2 to 6.2]
Statistical Analysis 7: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Social Functioning-SB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.1197, ANCOVA; Mean Difference (Final Values) = 2.8, 95% CI 2-sided [-0.7 to 6.4]
Statistical Analysis 8: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Social Functioning-DB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.2210, ANCOVA; Mean Difference (Final Values) = 2.1, 95% CI 2-sided [-1.3 to 5.5]
Statistical Analysis 9: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Role-Emotional-SB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.0847, ANCOVA; Mean Difference (Final Values) = 3.3, 95% CI 2-sided [-0.5 to 7.1]
Statistical Analysis 10: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Role-Emotional-DB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.0365, ANCOVA; Mean Difference (Final Values) = 4.0, 95% CI 2-sided [0.3 to 7.8]
Statistical Analysis 11: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Mental Health-SB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.2749, ANCOVA; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [-1.2 to 4.3]
Statistical Analysis 12: Comparison: Pregabalin CR DB vs Placebo DB; [analysis description as in outcome 11, analysis 11]; Test type: Superiority or Other; p = 0.0806, ANCOVA; Mean Difference (Final Values) = 2.5, 95% CI 2-sided [-0.3 to 5.2]
Statistical Analysis 13: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Physical component-SB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.0082, ANCOVA; Mean Difference (Final Values) = 2.0, 95% CI 2-sided [0.5 to 3.4]
Statistical Analysis 14: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Physical component-DB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.0008, ANCOVA; Mean Difference (Final Values) = 2.3, 95% CI 2-sided [1.0 to 3.7]
Statistical Analysis 15: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Mental component-SB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.2097, ANCOVA; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-0.8 to 2.5]
Statistical Analysis 16: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Mental component-DB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.1669, ANCOVA; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [-0.5 to 2.8]
Statistical Analysis 17: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Physical functioning-SB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.1466, ANCOVA; Mean Difference (Final Values) = 2.8, 95% CI 2-sided [-1.0 to 6.7]
Statistical Analysis 18: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Physical functioning-DB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.0439, ANCOVA; Mean Difference (Final Values) = 3.4, 95% CI 2-sided [0.1 to 6.7]
Statistical Analysis 19: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Role Physical-SB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.0250, ANCOVA; Mean Difference (Final Values) = 4.9, 95% CI 2-sided [0.6 to 9.3]
Statistical Analysis 20: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Role Physical-DB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.0107, ANCOVA; Mean Difference (Final Values) = 5.4, 95% CI 2-sided [1.3 to 9.5]

12. Secondary Outcome: Change in Mean Daily Sleep Interference Scores
Description: The pain related sleep interference item rating scale is scored on an 11 point numeric rating scale (NRS Sleep). It is self administered by the subject in order to rate how pain has interfered with their sleep during the past 24 hours, ranging from 0 (pain does not interfere with sleep) to 10 (completely interferes (unable to sleep due to pain)). Participants are to describe how their pain has interfered with their sleep during the past 24 hours by choosing the appropriate number on the numeric rating scale.
Time Frame: Week 19
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin CR DB | Placebo DB
Number analyzed (Participants) | 206 | 204
Units on a scale
  SB Baseline to Week 19 (N=205,203) | -4.5 (0.11) | -3.5 (0.11)
  DB Baseline to Week 19 (N=206,204) | -0.2 (0.10) | 0.7 (0.10)
Statistical Analysis 1: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for SB Baseline to Week 19.Estimates and p-values are from an analysis of covariance main effects model with baseline value, pooled center decided before unblinding, and treatment in the model; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.23 to -0.64]
Statistical Analysis 2: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for DB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with baseline value, pooled center decided before unblinding, and treatment in the model; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.12 to -0.58]

13. Secondary Outcome: Change in Hospital Anxiety and Depression Scales (HADS)
Description: The HADS is a self administered questionnaire that was designed to screen for the presence of a mood disorder in medically ill patients. To distinguish psychiatric presentations from physical illness, the items focus on subjective disturbance of mood rather than physical signs. The HADS contains 14 items rated on 4 point Likert type scales. Two subscales assess depression and anxiety. Each subscale consists of 7 statements, rated on a scale of 0 to 3 (0 = No anxiety or depression, to 3 = Severe feelings of anxiety or depression). Separate scores are calculated for each subscale ranging from 0 to 21. Higher scores denote greater severity of depression or anxiety
Time Frame: Week 19
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin CR DB | Placebo DB
Number analyzed (Participants) | 203 | 195
Units on a scale
  HADS-Anxiety-SB Baseline to Week 19 | -1.8 (0.21) | -1.1 (0.21)
  HADS-Anxiety-DB Baseline to Week 19 | 0.1 (0.19) | 0.9 (0.20)
  HADS-Depression-SB Baseline to Week 19 | -1.8 (0.20) | -1.2 (0.21)
  HADS-Depression-DB Baseline to Week 19 | 0.2 (0.19) | 0.8 (0.19)
Statistical Analysis 1: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for HADS-Anxiety-SB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.0154, ANCOVA; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.2 to -0.1]
Statistical Analysis 2: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for HADS-Anxiety-DB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.0027, ANCOVA; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.3 to -0.3]
Statistical Analysis 3: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for HADS-Depression-SB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.0166, ANCOVA; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.2 to -0.1]
Statistical Analysis 4: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for HADS-Depression-DB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p = 0.0217, ANCOVA; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.1 to -0.1]

14. Secondary Outcome: Change in the Brief Pain Inventory (BPI-sf)
Description: The BPI sf is a self-administered questionnaire developed to assess the severity of pain and the impact of pain on daily functions during a 24 hour period prior to evaluation. The BPI sf consists of 5 questions. Questions 1, 2, 3, and 4 measure pain on an 11 point scale from 0 (no pain) to 10 (worst pain possible). Question 5 consists of 7 item subsets which measure the level of interference of pain on daily functions on an 11 point scale from 0 (Does not interfere) to 10 (Completely interferes).
Time Frame: Week 19
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin CR DB | Placebo DB
Number analyzed (Participants) | 203 | 195
Units on a scale
  Pain Severity Index-SB Baseline to Week 19 | -18.0 (0.47) | -13.8 (0.49)
  Pain Severity Index-DB Baseline to Week 19 | -0.7 (0.43) | 3.1 (0.44)
  Pain Interference Index-SB Baseline to Week 19 | -21.9 (0.71) | -17.2 (0.74)
  Pain Interference Index-DB Baseline to Week 19 | -0.2 (0.67) | 4.0 (0.70)
Statistical Analysis 1: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Pain Severity Index-SB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -4.2, 95% CI 2-sided [-5.5 to -3.0]
Statistical Analysis 2: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Pain Severity Index-DB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -3.8, 95% CI 2-sided [-5.0 to -2.7]
Statistical Analysis 3: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Pain Interference Index-SB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -4.6, 95% CI 2-sided [-6.5 to -2.7]
Statistical Analysis 4: Comparison: Pregabalin CR DB vs Placebo DB; This ANCOVA model analysis is for Pain Interference Index-DB Baseline to Week 19. Estimates and p-values are from an analysis of covariance main effects model with SB baseline value, center, and treatment in the model; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -4.2, 95% CI 2-sided [-6.0 to -2.4]

15. Secondary Outcome: Percentage of Participants With Benefit From Treatment, Satisfaction With Treatment and Willingness to Continue Treatement (BSW)
Description: The BSW is administered by the study physician or designated site personnel and consists of three single item measures designed to capture the patient's perception of the effect of treatment in terms of the relative benefit, their satisfaction, and their intention or willingness to continue on therapy.
Time Frame: Week 19
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin CR DB | Placebo DB
Number analyzed (Participants) | 201 | 193
Percentage of participants
  Benefit from treatment | 98.5 | 93.3
  Satisfaction with treatment | 96.0 | 90.7
  Willingness to continue treatment | 87.6 | 81.3
Statistical Analysis 1: Comparison: Pregabalin CR DB vs Placebo DB; This analysis is for 'Benefit from treatment'. Proportional odds logistic regression was used with a term for treatment in the model; Test type: Superiority or Other; p = 0.0161, Regression, Logistic; Odds Ratio (OR) = 4.77, 95% CI 2-sided [1.34 to 17.00] — Odds ratio was the probability of the event occurring in pregabalin CR DB relative to the event occurring in placebo DB. Odds ratio > 1 was in favor of pregabalin CR
Statistical Analysis 2: Comparison: Pregabalin CR DB vs Placebo DB; This analysis is for 'Satisfaction with treatment'. Proportional odds logistic regression was used with a term for treatment in the model; Test type: Superiority or Other; p = 0.0378, Regression, Logistic; Odds Ratio (OR) = 2.48, 95% CI 2-sided [1.05 to 5.85] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 3: Comparison: Pregabalin CR DB vs Placebo DB; This analysis is for 'Willingness to continue treatment'. Proportional odds logistic regression was used with a term for treatment in the model; Test type: Superiority or Other; p = 0.0901, Regression, Logistic; Odds Ratio (OR) = 1.61, 95% CI 2-sided [0.93 to 2.81] — [estimate comment as in outcome 15, analysis 1]

16. Secondary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. A serious adverse event is any untoward medical occurrence at any dose that: Results in death; Is life-threatening (immediate risk of death); Requires inpatient hospitalization or prolongation of existing hospitalization; Results in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); or Results in congenital anomaly/birth defect. The study physician used the adjective "severe" to those AEs that interfere significantly with participant's usual function.
Time Frame: Baseline to Week 20
Population: The SB Analysis Set (SBAS) consisted of all participants who were enrolled into the SB phase of the study and received at least 1 dose of study medication; The FAS consisted of all participants randomized to the DB phase who received at least 1 dose of study medication in the DB phase.
  Both SBAS and FAS were included in this analysis.
Measure: Number; unit: Participants
Arm/Group | Pregabalin CR DB | Placebo DB | Pregabalin CR SB
Number analyzed (Participants) | 208 | 205 | 801
Participants
  Participants with AEs | 80 | 63 | 441
  Participants with Serious AEs | 7 | 3 | 17
  Participants with Severe AEs | 9 | 3 | 35

17. Secondary Outcome: Percentage of Participants With Suicidal Behaviour/Ideation
Description: Percentage of participants with suicidal behavior/ideation were noted as Baseline, Weeks 6, 11, 15, 19 and 20.
Time Frame: Baseline, Weeks 6, 11, 15, 19 and 20
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin CR DB | Placebo DB
Number analyzed (Participants) | 208 | 205
Percentage of participants
  SB BL(N=208,205) | 0 | 0.5
  Week 6 (N=208,205) | 0 | 0
  Week 11 (N=194,178) | 0 | 0
  Week 15 (N=183,167) | 0 | 0
  Week 19 (N=204,197) | 0 | 0
  Week 20 (N=199,194) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to Week 20
Description: The SB analysis set (SBAS) consisted of all participants who were enrolled into the SB phase of the study and received at least 1 dose of study medication; The FAS consisted of all participants randomized to the DB phase who received at least 1 dose of study medication in the DB phase. Both SBAS and FAS were included in this analysis
Arm/Group | Pregabalin CR DB | Placebo DB | Pregabalin CR SB
Serious Adverse Events (participants affected / at risk) | 7/208 | 3/205 | 17/801
Other Adverse Events (participants affected / at risk) | 7/208 | 1/205 | 202/801
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin CR DB (N=208) | Placebo DB (N=205) | Pregabalin CR SB (N=801)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular disorder (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Renal mass (Renal and urinary disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sexual abuse (Social circumstances) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin CR DB (N=208) | Placebo DB (N=205) | Pregabalin CR SB (N=801)
Dizziness (Nervous system disorders) | 7 | 1 | 137
Somnolence (Nervous system disorders) | 1 | 0 | 91

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.